CLINICAL TRIAL: NCT03467113
Title: An Open-Label Trial to Assess the Safety of ZX008 (Fenfluramine Hydrochloride) Oral Solution in Combination With Cannabidiol, as an Adjunctive Therapy in Children and Young Adults With Dravet Syndrome or Lennox-Gastaut Syndrome
Brief Title: A Study to Assess the Safety and Tolerability of ZX008 in Children and Young Adults With Dravet Syndrome or Lennox Gastaut Syndrome Currently Taking Cannabidiol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zogenix International Limited, Inc., a subsidiary of Zogenix, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZX008-1602
Record Dates: First submitted 2018-01-30; First posted 2018-03-15 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Dravet Syndrome; Lennox Gastaut Syndrome
Keywords: Dravet Syndrome; LGS
MeSH Terms: conditions — Epilepsies, Myoclonic; Lennox Gastaut Syndrome | interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ZX008 0.2 to 0.8 mg/kg/day (Experimental): ZX008 is supplied as an oral solution in a concentration of 2.5 mg/mL. Subjects will receive open-label ZX008 (flexible dosing 0.2 mg/kg/day to 0.8 mg/kg/day)
  Interventions: Drug: ZX008 0.2 to 0.8 mg/kg/day; Drug: Cannabidiol

INTERVENTIONS:
Drug: ZX008 0.2 to 0.8 mg/kg/day — ZX008 drug is an oral aqueous solution of fenfluramine hydrochloride. The product is sugar free.
Drug: Cannabidiol — Cannabidiol

SUMMARY:
This is an open label study to evaluate the safety of ZX008 (fenfluramine) in patients with Dravet syndrome (DS) or Lennox Gastaut syndrome (LGS) who are being administered cannabidiol (CBD).

ELIGIBILITY:
Key Inclusion Criteria:

* Subject has a clinical diagnosis of DS or LGS, where convulsive seizures (generalized tonic clonic seizures, tonic seizures, atonic seizures, tonic/atonic seizures, focal seizures with clear observable motor signs) are not completely controlled by current AEDs.
* All medications or interventions for epilepsy (including ketogenic diet [KD] and vagal nerve stimulation [VNS]) must be stable for at least 4 weeks prior to first ZX008 dose and are expected to remain stable throughout the study.
* Subjects must be taking a stable dose of CBD for at least 4 weeks prior to first ZX008 dose.
* Subject's source of CBD is expected to be consistent for at least 3 months during study participation.

Key Exclusion Criteria:

* Subject has current or past history of cardiovascular or cerebrovascular disease, myocardial infarction or stroke.
* Subject with current cardiac valvulopathy or pulmonary hypertension that the Investigator, parent/caregiver, Independent Cardiac Advisory Board, Independent Data and Safety Monitoring Committee, or sponsor deems clinically significant.
* Subject has a current or past history of glaucoma.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2020-06-24 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Baseline to Day 365
  Number of adverse events including serious adverse events, number of adverse events leading to study withdrawal
Change in Heart Rate | Baseline to Day 365
  Change in resting heart rate using standard measures
Change in blood pressure | Baseline to Day 365
  Change in resting blood pressure using standard measures
Change in temperature | Baseline to Day 365
  Change in resting temperature using standard measures
Change in respiratory rate | Baseline to Day 365
  Change in resting respiratory rate using standard measures
Changes in heart rhythm | Baseline to Day 365
  Changes in heart beat as measured with 12-lead electrocardiogram
Changes in heart valve function | Baseline to Day 365
  Changes in heart valves as measured with standard echocardiogram
Changes in treatment-emergent body weight and height | Baseline to Day 365
  Changes in body weight and height by report of BMI in kg/m^2

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - PANDA Neurology/CIRCA, Atlanta, Georgia
  - MultiCare Institute for Research & Innovation, Tacoma, Washington